CLINICAL TRIAL: NCT04484571
Title: Robotic Rehabilitation and Multimodal Instrumented Assessment of Post-stroke Elbow Motor Functions - a Randomized Controlled Trial Protocol
Brief Title: Multimodal Instrumented Assessment of Post-stroke Elbow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Azienda USL Toscana Nord Ovest (Other)
Collaborators: Scuola Superiore Sant'Anna Pisa (Unknown)
Responsible Party: Principal Investigator, Federico Posteraro, Head of North Area Rehabilitation Department, Azienda USL Toscana Nord Ovest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEEM20160118
Record Dates: First submitted 2020-07-10; First posted 2020-07-23 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Spasticity, Muscle; Stroke; Upper Limb
Keywords: Robotics; Upper extremities; EMG
MeSH Terms: conditions — Muscle Spasticity; Stroke

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Outcomes Assessor
Masking Description: Indipendent assessor blinded on treatment provided
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic treatment (Experimental): Patients receive 4 weeks of elbow rehabilitation treatment provided by the NEEM robotic elbow exoskeleton
  Interventions: Device: Neuroexsos elbow module
- Conventional treatment (Active Comparator): Patients receive 4 weeks of elbow conventional rehabilitation treatment matched in time
  Interventions: Device: Neuroexsos elbow module

INTERVENTIONS:
Device: Neuroexsos elbow module — The treatment group will be further divided into two levels (sub-groups), based on pathological severity: Level 1 corresponds to an FM score equal or below 28, and Level 2 with FM greater than 28. The two sub-groups will receive different combinations of robotically assisted passive mobilization (PM) and active mobilization (AM) treatment modalities, according to their differing clinical needs

SUMMARY:
The proposed clinical trial will employ the NEUROExos Elbow Module (NEEM), an active robotic exoskeleton, for the passive mobilization and active training of elbow flexion and extension in 60 sub-acute and chronic stroke patients with motor impairments (hemiparesis and/or spasticity) of the right arm. The study protocol is a randomized controlled trial consisting of a 4-week functional rehabilitation program, with both clinical and robotically instrumented assessments to be conducted at baseline and post-treatment.

DETAILED DESCRIPTION:
The reliable assessment, attribution, and alleviation of upper-limb joint stiffness are essential clinical objectives in the early rehabilitation from stroke and other neurological disorders, to prevent the progression of neuromuscular pathology and enable proactive physiotherapy towards functional recovery. However, the current clinical evaluation and treatment of this stiffness (and underlying muscle spasticity) are severely limited by their dependence on subjective evaluation and manual limb mobilization, thus rendering the evaluation imprecise and the treatment insufficiently tailored to the specific pathologies and residual capabilities of individual patients. To address these needs, the proposed clinical trial will employ the NEUROExos Elbow Module (NEEM), an active robotic exoskeleton, for the passive mobilization and active training of elbow flexion and extension in stroke patients with motor impairments (hemiparesis and/or spasticity) of the right arm. The study protocol provide a functional rehabilitation program, with both clinical and robotically instrumented assessments to be conducted at baseline and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Upper limb spasticity due to neurological impairment;
* Cognitive abilities sufficient for understanding instructions;
* Absence of severe pain assessed as Visual Analogic Score (VAS) < 4 (range 0-10).

Exclusion Criteria:

* Unstable general clinical conditions;
* Inability to keep sitting posture;
* Tendon retractions limiting upper limb joints range of motion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in the score of the upper-extremity section of Fugl-Meyer assessment scale (FM 0-66) higher score means better | before and within 1 week after 4 weeks of treatment
  It is a clinical scale used for the assessment of motor function in stroke patients
Change in the score of Modified Ashworth Scale (MAS 0-5 scoring 1+ as 2 for statistical analysis) higher score means worse | Before and within 1 week after 4 weeks of treatment
  It is a clinical scale for spasticity assessment

SECONDARY OUTCOMES:
Change in Maximum Extension Torque (MET) | Before and within 1 week after 4 weeks of treatment
  It corresponds to the maximum torque value recorded during a static hold phase at the maximum reached extension angle
Change in Zero Torque Angle (ZTA) | Before and within 1 week after 4 weeks of treatment
  It is the angular value corresponding to null torque exerted by the robot; in this configuration, flexor and extensor torques are equal and opposite and the system is ideally not applying any force to hold the elbow in position, which has reached its equilibrium point
Change in Joint Impedance (JIMP) | Before and within 1 week after 4 weeks of treatment
  A measure of the limb resistance to muscle elongation, extracted as the ratio between joint torque and joint angular position for constant, slow-speed movements, the main contribution to the joint impedance can be identified in the joint stiffness (i.e. rigidity).

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Versilia, Camaiore, Lucca, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pilla A, Trigili E, McKinney Z, Fanciullacci C, Malasoma C, Posteraro F, Crea S, Vitiello N. Robotic Rehabilitation and Multimodal Instrumented Assessment of Post-stroke Elbow Motor Functions-A Randomized Controlled Trial Protocol. Front Neurol. 2020 Oct 22;11:587293. doi: 10.3389/fneur.2020.587293. eCollection 2020. PMID 33193052